CLINICAL TRIAL: NCT05686902
Title: Comparison of Two Different Solutions for Peristomal Skin Care in Patients With Pediatric Stoma: A Randomized Controlled Clinical Study
Brief Title: Comparison of Two Different Solutions for Peristomal Skin Care in Patients With Pediatric Stoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, ESRA ARDAHAN AKGUL, Assistant Professor, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 781
Record Dates: First submitted 2022-12-30; First posted 2023-01-17 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Colostomy Site

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PH 5.5 BABY SHAMPOO GROUP (Experimental): Distilled water+Ph 5.5 baby shampoo for stoma care of patients in the first group
  Interventions: Other: CLEANING SOLUTION
- SERUM PHYSIOLOGIC GROUP (Active Comparator): 0.9% saline solution for stoma care of patients in the second group
  Interventions: Other: CLEANING SOLUTION

INTERVENTIONS:
Other: CLEANING SOLUTION — The difference in peristomal skin integrity between the groups will be examined.

SUMMARY:
The aim of this study is to determine the effect of two different skin care solutions used in stoma care on peristomal skin integrity and compare them with each other.

DETAILED DESCRIPTION:
ABSTRACT

The research was planned as a randomized controlled experiment. Simple stratified randomization according to age will be done. The purpose of the study will be explained to the children and their parents who agreed to participate in the study and their consent will be obtained.

Study Groups: In the study, there will be 2 groups with 12 patients in each group.

* Distilled water+Ph 5.5 baby shampoo for stoma care of patients in the first group (routine care of the clinic)
* 0.9% saline solution for stoma care of patients in the second group Randomization: It will be provided as 2 groups, using the Random Sequence Generator on www.random.org. The randomization provided by the program can be accessed from the link https://www.random.org/integers/?num=24&min=1&max=24&col=2&base=10&format=html&rnd=new.

Intervention Procedure: After obtaining written consent, peristomal skin integrity of all participants will be evaluated on day 0 post-op prior to randomization.

Peristomal Skin Integrity Assessment:

* Stoma circumference skin pH measurement
* Skin temperature measurement around stoma
* Measurement of skin moisture around the soma
* Pittman Ostomy Complication Severity Index measurement (It is a 9-parameter evaluation scale developed by Joyce Pittman in 2014, and its validity and reliability in Turkish were performed by Arslantaş et al. in 2019. The purpose of the scale is to evaluate the frequency and severity of early postoperative complications during follow-up in individuals with stoma. This index Evaluates leakage, peristomal irritant dermatitis, pain, bleeding in or around the stoma, stomal necrosis, stenosis, retraction, mucocutaneous separation, and hyperplasia All complications 0 to 3 (0 = absent, 1 = mild, 2 = moderate, 3 = severe) (The total score ranges from 0 to 27. Higher scores indicate more severe ostomy complications) Between the 0th and 7th day following the stoma opening, stoma care will be applied to the patients by the same researcher every day, through the skin care solution specific to the group they are in. Peristomal skin integrity of the patients will be evaluated on the 3rd and 7th days of the study. Only children who can be observed from day 0 following stoma opening and whose stoma can be cared for for at least 7 days will be included in the study. The skin pH value around the stoma will be evaluated with the BRD Digital Ph Meter, the temperature measurement will be evaluated with the infrared thermometer used routinely in the clinic, and the humidity measurement will be evaluated with the BRD Digital Skin Moisture Analyzer.

Statistical Analysis: A researcher who does not know which group the patients are in will perform the statistical analysis of the study using the single-blind method. Analysis of the data obtained from the research will be carried out in IBM® SPSS Statistics Version 22 program. Age, gender, etc. of the patients in the study. demographic characteristics will be given as number and percentage distributions. Comparisons of numerical variables between groups; It will be evaluated with a non-parametric or parametric appropriate test by looking whether the normal distribution condition is met. In the study, the statistical significance value was determined as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients who volunteered to participate in the study and received Informed Voluntary Consent from their parents.
* Products used in routine clinical care in skin care (distilled water + baby shampoo), patients for whom the use of 0.9% saline is appropriate
* Patients who do not have any other underlying disease that may affect peristomal skin integrity
* Patients included in the study from the 0th day following the colostomy opening
* Patients who can be observed at least on the 7th day

Exclusion Criteria:

* Patients who did not volunteer to participate in the study and who could not obtain Informed Voluntary Consent from their parents
* Patients with a stoma other than a colostomy (ileostomy, etc.)
* Products used in routine clinical care in skin care (distilled water + baby shampoo), patients for whom the use of 0.9% saline is not suitable
* Patients with another underlying disease that may affect peristomal skin integrity
* Patients on the 1st day and after the colostomy opening
* Patients who cannot be observed for at least 7 days

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
skin pH measurement around stoma | change between the 0th and the 7th day
  skin pH measurement around stoma will be measured with a portable device brand BRD
Skin temperature measurement around stoma | change between the 0th and the 7th day
  Skin temperature measurement around stoma will be measured with a portable infrared device.
skin moisture around the soma | change between the 0th and the 7th day
  percent of (%)skin moisture around the soma will be measured with a portable device brand BRD
Pittman Ostomy Complication Severity Index | change between the 0th and the 7th day
  It is a 9-parameter evaluation scale developed by Joyce Pittman in 2014, and its validity and reliability in Turkish were performed by Arslantaş et al. in 2019. The purpose of the scale is to evaluate the frequency and severity of early postoperative complications during follow-up in individuals with stoma. This index Evaluates leakage, peristomal irritant dermatitis, pain, bleeding in or around the stoma, stomal necrosis, stenosis, retraction, mucocutaneous separation, and hyperplasia All complications 0 to 3 (0 = absent, 1 = mild, 2 = moderate, 3 = severe) (The total score ranges from 0 to 27. Higher scores indicate more severe ostomy complications)

CONTACTS AND LOCATIONS:
Overall Officials: Esra ARDAHAN AKGÜL, Asst. Prof., Principal Investigator — İzmir Katip Çelebi University
Locations (1):
- Behçet Uz Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No